CLINICAL TRIAL: NCT01756105
Title: Gestational Diabetes in Non Obese Women and Metformine
Brief Title: Efficacy of Metformin in Achieving Glycaemia Goals as Recommended for the Treatment of Gestational Diabetes in Non Obese Women
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4965
Record Dates: First submitted 2012-12-19; First posted 2012-12-24 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Gestational Diabetes; Metformin; Treatment; Oxidative Stress
MeSH Terms: conditions — Diabetes, Gestational | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- treatment by Metformin plus insulin if needed (Experimental): Metformin: from 500 mg 2 time per day to 2500 mg per day; with increment of 500 mg every 5 days until abstention of
  Interventions: Drug: Metformin; Drug: Rapid acting analog insulin Intermediate acting NPH Insulin
- treatment by insulin (Active Comparator): Insulin therapy:If post meal (2 hours after meal) glycaemia is > to 120 mg/dl introduce Insulin rapid acting analog (Humalog*, Novorapid*) before the meal concerned and according to the weight. If weight is < 80 kg: breakfast 5U, lunch time 3U, and dinner 4U. If weight is > 80 kg :breakast 6U, lunch time 4U, dinner 5U.If post meal glycaemia stay over 120 mg/dl but lower than130 mg/dl: do 1 U more.If post meal glycaemia stay over 140 mg/dl : do 2 UI moreIf fasting glycaemia is over 95 mg/dl : introduce NPH Insulin (Umuline NPH*, insulatard*) before sleeping : 5U if weight is < 80 kg - 6U if weight is > 80 kgIf fasting glycaemia stay over 95 mg/dl increase NPH Insulin for 1 U and for 2 U if fasting glycaemia is over 110 mg/dl.
  Interventions: Drug: Rapid acting analog insulin Intermediate acting NPH Insulin

INTERVENTIONS:
Drug: Metformin — Metformin: from 500 mg 2 time per day to 2500 mg per day; with increment of 500 mg every 5 days until abstention of
  Arms: treatment by Metformin plus insulin if needed
Drug: Rapid acting analog insulin Intermediate acting NPH Insulin — Insulin therapy:If post meal (2 hours after meal) glycaemia is > to 120 mg/dl introduce Insulin rapid acting analog (Humalog*, Novorapid*) before the meal concerned and according to the weight. If weight is < 80 kg: breakfast 5U, lunch time 3U, and dinner 4U. If weight is > 80 kg :breakast 6U, lunch time 4U, dinner 5U.If post meal glycaemia stay over 120 mg/dl but lower than130 mg/dl: do 1 U more.If post meal glycaemia stay over 140 mg/dl : do 2 UI moreIf fasting glycaemia is over 95 mg/dl : introduce NPH Insulin (Umuline NPH*, insulatard*) before sleeping : 5U if weight is < 80 kg - 6U if weight is > 80 kgIf fasting glycaemia stay over 95 mg/dl increase NPH Insulin for 1 U and for 2 U if fasting glycaemia is over 110 mg/dl.

SUMMARY:
Gestational diabetes (GD) is defined by a hyperglycemia discovered during pregnancy, leading to fetal and maternal complications which may be prevented by reaching very strict glycaemia targets. Prevalence depends on patient's ethnic group and is about 6 to 14%. This prevalence is increasing due to increased GD risk factors (obesity, pregnancy over 35) and also because criteria of screening have been strengthened after the results of last studies. Usual treatment is diet and in case of failure insulin therapy with multiple injections which may lead to hypoglycemia and weight gain and is very difficult to manage for patients. Some studies have shown the comparable effect of metformin and insulin in about 50% of GD obese patients. The aim of our study is to evaluate efficacy of metformin, outcomes in mother and fetus and baby of metformin. In case of metformin failure, insulin will be added in order to obtain glycaemia in desired goals.Oxidative stress will be assessed in mother blood, baby umbilical cord blood, baby umbilical cord and placenta in 90 women and the oxidative stress compared between insulin and metformin alone treated patients.

ELIGIBILITY:
Inclusion Criteria:

Women.

* Age more than 18 and less than 40 years.
* Unique spontaneous pregnancy.-BMI less than 30kg/m2 before pregnancy.
* 24 to 30 weeks of amenorrhea or 22 to 28 weeks of gestation.
* Gestational diabetes.
* Social Security affiliated subject.- Patient able to understand and signed informed consent.

Exclusion Criteria:

* Contraindications to metformin.
* Metformin treatment prior to protocol inclusion.
* Multiple pregnancies.
* Diabetes diagnosed prior to pregnancy.
* High blood pressure prior to pregnancy.
* Pregnancy hepatic complication
* High blood pressure prior to study inclusion.
* Pre or eclampsia.- Premature membranes rupture.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2012-06 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Efficacy of metformin in treatment of gestational diabetes based on capillary glycaemia with an objective of less than 6 measures out of range | After diagnosis of gestational diabetes and until 3 months after delivery; screening made between 22th and 28th week of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Jeandidier, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (5):
- France (5):
  - Hôpitaux Civils de Colmar, Colmar
  - CHU Dijon,, Dijon
  - Centre hospitalier de Mulhouse, Mulhouse
  - CHU de Reims, Reims
  - Hôpitaux Universitaires de Strasbourg, Strasbourg